CLINICAL TRIAL: NCT00151658
Title: Randomized Multicenter Comparison of Sirolimus Versus Bare Metal Stent Implantation in Complex Coronary Lesions. Acronym: Scand Stent
Brief Title: Sirolimus Eluting Stents in Complex Coronary Lesions (SCANDSTENT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCANDSTENT
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Ischaemic Heart Disease
Keywords: Coronary complex lesions; Restenosis; Drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Coronary Drug Eluting Stents for PCI

SUMMARY:
The purpose of this study is to evaluate the clinical and angiographic outcome of implantation of stents eluting or not eluting Sirolimus in patients with complex coronary artery lesions suitable for percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

Stable, or unstable angina and/or objective signs of myocardial ischaemia Lesions should be de novo and located in native vessels with a diameter > 2.25 mm.

Complex lesions to be included should have at least one of the following characteristics:

* Ostial in location (< 5 mm from ostium)
* Total occlusions with a length ≥ 15 mm
* Bifurcational (side branch > 1.75 mm in diameter)
* Angulated (> 45° within lesion)

Exclusion Criteria:

Patients:

* Other severe disease with an expected survival < 1 year
* Other significant cardiac disease
* Known allergy against paclitaxel, clopidogrel or stainless steel.
* Myocardial infarction within 3 days of the index procedure
* Linguistic difficulties needing an interpreter
* Renal insufficiency (p-creatinine > 200 micromol/l)
* Gastrointestinal bleeding within 1 month
* Childbearing potential or pregnancy
* Participation in another study

Lesions:

* Unprotected left main disease
* Restenosis
* Lesions containing visible thrombus
* Treatment with other modality than balloon or stent (ablation, brachytherapy, ultrasound) in connection with the index procedure
* Diffuse coronary disease distal to the treated lesion
* Heavily calcification
* Lesion located in saphenous vein graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322
Dates: Start 2002-10; Study Completion 2006-06

PRIMARY OUTCOMES:
Minimal lumen diameter
Frequency of restenosis (>50%) at 6 months.

SECONDARY OUTCOMES:
Diameter stenosis, late loss and loss index at 6 months MACE: death, myocardial infarction, target lesion revascularisation within 12 months and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Henning Kelbaek, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Kelbaek H, Klovgaard L, Helqvist S, Lassen JF, Krusell LR, Engstrom T, Botker HE, Jorgensen E, Saunamaki K, Aljabbari S, Thayssen P, Galloe A, Jensen GV, Thuesen L. Long-term outcome in patients treated with sirolimus-eluting stents in complex coronary artery lesions: 3-year results of the SCANDSTENT (Stenting Coronary Arteries in Non-Stress/Benestent Disease) trial. J Am Coll Cardiol. 2008 May 27;51(21):2011-6. doi: 10.1016/j.jacc.2008.01.056. PMID 18498953